CLINICAL TRIAL: NCT00008463
Title: A Prospective, Multicenter, Phase II/III, Open-Label, Controlled, Randomized Trial Evaluating the Efficacy, Safety, and Tolerability of Interferon-alfa-2a Plus Ribavirin Versus PEG-interferon-alfa-2a Plus Ribavirin for Chronic Hepatitis C Virus (HCV) Infection in Individuals Co-Infected With Human Immunodeficiency Virus-1 (HIV-1)
Brief Title: A Comparison of the Effectiveness, Safety, and Tolerability of Two Different Hepatitis C Treatments in Patients Infected With Both HIV and Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5071; 10675 (Registry Identifier: DAIDS ES Registry Number); Substudy AACTG A5091s; ACTG A5071; AACTG A5071
Record Dates: First submitted 2001-01-09; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Ribavirin; Polyethylene Glycols; Interferon Alfa-2a; HIV-1; Antiviral Agents; Hepatitis C, Chronic
MeSH Terms: conditions — HIV Infections; Hepatitis C; Hepatitis C, Chronic | interventions — Ribavirin; Interferon alpha-2; peginterferon alfa-2a

INTERVENTIONS:
Drug: Ribavirin
Drug: Interferon alfa-2a
Drug: Peginterferon alfa-2a

SUMMARY:
The purpose of this study is to see if treatment with PEG-interferon-alfa-2a (PEG-IFN) plus ribavirin is a more effective treatment for hepatitis C virus (HCV) than interferon-alfa-2a (IFN) plus ribavirin for patients infected with both HCV and HIV. The study will also compare the 2 regimens to see which has fewer side effects.

HCV infection is common in patients infected with HIV. Patients infected with both HIV and HCV viruses seem to have more severe hepatitis C. A combination of IFN and ribavirin has been shown to lessen the severity of HCV. PEG-IFN is a modified form of IFN that stays in the blood longer, which means that patients would not have to take the treatment as often. This study will compare the safety and effectiveness of PEG-IFN to IFN when each is combined with ribavirin.

DETAILED DESCRIPTION:
Infection with HCV is common in patients infected with HIV owing to similar routes of transmission. The cellular immunosuppression caused by HIV infection appears to lead to an increased HCV plasma load, more progressive liver disease, and, in patients with chronic hepatitis C, increased mortality. Ribavirin treatment combined with IFN has shown improved sustained virologic response rates over IFN monotherapy. PEG-IFN, a chemically modified formulation of IFN, circulates for a much longer time in the blood than the parent compound. Pharmacokinetic and pharmacodynamic data suggest that PEG-IFN injected weekly would have the potential for superior efficacy as compared with IFN injected 3 times per week. The efficacy and safety profiles of combination therapy with PEG-IFN and ribavirin are not well known. This study will compare combination therapy consisting of PEG-IFN and ribavirin with that of IFN and ribavirin.

Patients are stratified according to HCV genotype and CD4 count and viral load, then randomized to either Arm A (IFN plus ribavirin) or Arm B (PEG-IFN plus ribavirin). Patients receive up to 48 weeks of treatment. Virologic response is assessed at Week 24 and a decision to continue or discontinue treatment is made. If a virologic response is shown at Week 24, the patient continues treatment for an additional 24 weeks. If no virologic response is observed, then the histologic response is assessed by a liver biopsy. If biopsy shows a histologic response is present, treatment is continued for 24 weeks. If biopsy shows no histologic response, treatment is discontinued. [AS PER AMENDMENT 07/20/01: Patients with virologic response who discontinue after Week 24 will have liver biopsy at time of discontinuation. Patients with no virologic response continuing study treatment after having a liver biopsy within 2 weeks of Week 24, who also demonstrate histologic response and decide to discontinue after Week 24, are strongly encouraged to have a 2nd liver biopsy at the end of treatment. Patients with no virologic response who discontinue after Week 24 will not have liver biopsy at time of discontinuation.] Physical examinations are done regularly and blood samples collected for routine laboratory tests, confidential genetic testing, and to measure HCV and HIV-1 plasma viral loads. Women able to become pregnant have regular pregnancy tests. All patients are followed for an additional 24 weeks after treatment discontinuation.

Patients may enroll in 1 or none of the following substudies: A5091s, Hepatic C Viral Kinetics in Subjects Co-infected with Human Immunodeficiency Virus-1 (HIV-1) and Hepatitis C Virus Genotype 1 (HCV-1); [AS PER AMENDMENT 07/20/01: The following text has been deleted: or A5092s, Evaluation of the Effects of Ribavirin on Zidovudine (ZDV) or Stavudine (d4T) Triphosphate Formation] [AS PER AMENDMENT 07/20/01: Substudy A5092s, Evaluation of the Effects of Ribavirin on Zidovudine (ZDV) or Stavudine (d4T) Triphosphate Formation is now a stand-alone study.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have chronic liver disease consistent with chronic hepatitis C.
* Have evidence of hepatitis C within the 48 weeks prior to entry.
* Are 18 to 65 years old.
* Agree to use 2 barrier methods of birth control during the study and for 6 months after stopping the medications.
* Meet 1 of the following sets of guidelines: 1) have a CD4 count of more than 100 cells/mm3 and have a viral load (level of HIV in the blood) of less than 10,000 copies/ml within 35 days prior to study entry, and have taken stable anti-HIV drugs for at least 12 weeks prior to study entry and plan to remain on the same treatment for the first 24 weeks of the study; or 2) have a CD4 count of more than 300 cells/mm3 within 35 days prior to study entry and have not taken any anti-HIV drugs in the 12 weeks prior to entry, and do not plan to start anti-HIV treatment within the first 24 weeks of study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a positive test for hepatitis B.
* Show evidence of medical conditions associated with long-term liver disease other than HCV.
* Have severe mental illness, especially depression, or have been hospitalized for mental illness within the previous 24 weeks.
* Are allergic to any of the study products.
* Have uncontrolled seizures.
* Have had or currently have any immune diseases.
* Have lung disease such that function is limited.
* Have had evidence of heart disease or certain heart problems within 24 weeks of study entry.
* Have severe retinopathy (eye disease).
* Have had a major organ transplant and still have the graft.
* Have any other severe disease or cancer that would interfere with the study.
* Have had anti-cancer or immune-regulating drugs or radiation treatment within 24 weeks of study entry or expect to need such treatment during the study.
* Have received rifampin, rifabutin, pyrazinamide, isoniazid, ganciclovir, hydroxyurea, granulocyte colony-stimulating factor (G-CSF), or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 6 weeks of study entry.
* Abuse drugs or alcohol. Patients in methadone programs may participate.
* Have a blood disorder such as thalassemia.
* Have received interferon or oral ribavirin therapy.
* Have taken an experimental drug that affects HCV, within 6 weeks of study entry.
* Need to use during the study any of the drugs prohibited by the study.
* Have had an opportunistic (AIDS-related) infection within 4 weeks of study entry.
* Are pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2000-11; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Study Chair — Harvard/Massachusetts General Hospital; Paul Volberding, MD, Study Chair — San Francisco General Hospital
Locations (24):
- United States (24):
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Mt. Sinai Med. Ctr. A0404 CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - AIDS Care CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Philadelphia Veterans Admin. Med. Ctr. A6205 CRS, Philadelphia, Pennsylvania
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas

REFERENCES:
- [Result] R Chung, J Andersen, P Volberding, G Robbins, T Liu, K Sherman, M Peters, M Koziel, B Alston, D Colquhoun, T Nevin, G Harb, C van der Horst, and AIDS Clinical Trials Group A5071 Study Team: A Randomized, Controlled Trial of PEG-Interferon-alfa-2a plus Ribavirin vs Interferon-alfa-2a plus Ribavirin for Chronic Hepatitis C Virus Infection in HIV-co-infected Persons: Follow-up Results of ACTG A5071. CROI 2004. Abstract 110.
- [Result] Chung RT, Andersen J, Volberding P, Robbins GK, Liu T, Sherman KE, Peters MG, Koziel MJ, Bhan AK, Alston B, Colquhoun D, Nevin T, Harb G, van der Horst C; AIDS Clinical Trials Group A5071 Study Team. Peginterferon Alfa-2a plus ribavirin versus interferon alfa-2a plus ribavirin for chronic hepatitis C in HIV-coinfected persons. N Engl J Med. 2004 Jul 29;351(5):451-9. doi: 10.1056/NEJMoa032653. PMID 15282352
- [Result] Plosker GL, Keating GM. Peginterferon-alpha-2a (40kD) plus ribavirin: a review of its use in hepatitis C Virus And HIV co-infection. Drugs. 2004;64(24):2823-43. doi: 10.2165/00003495-200464240-00009. PMID 15563253
- [Result] Sherman KE, Shire NJ, Rouster SD, Peters MG, James Koziel M, Chung RT, Horn PS. Viral kinetics in hepatitis C or hepatitis C/human immunodeficiency virus-infected patients. Gastroenterology. 2005 Feb;128(2):313-27. doi: 10.1053/j.gastro.2004.11.059. PMID 15685543
- [Result] Graham CS, Wells A, Liu T, Sherman KE, Peters M, Chung RT, Bhan AK, Andersen J, Koziel MJ; ACTG 5071 Study Team. Antigen-specific immune responses and liver histology in HIV and hepatitis C coinfection. AIDS. 2005 May 20;19(8):767-73. doi: 10.1097/01.aids.0000168970.80551.3d. PMID 15867490
- [Result] Jones R, Dunning J, Nelson M. HIV and hepatitis C co-infection. Int J Clin Pract. 2005 Sep;59(9):1082-7. doi: 10.1111/j.1742-1241.2005.00596.x. PMID 16115185
- [Result] Graham CS, Wells A, Liu T, Sherman KE, Peters M, Chung RT, Bhan AK, Andersen J, Koziel MJ; ACTG 5071 Study Team. Relationships between cellular immune responses and treatment outcomes with interferon and ribavirin in HIV/hepatitis C virus co-infection. AIDS. 2006 Feb 14;20(3):345-51. doi: 10.1097/01.aids.0000206500.16783.2e. PMID 16439867
- [Result] Bhattacharya D, Umbleja T, Carrat F, Chung RT, Peters MG, Torriani F, Andersen J, Currier JS. Women experience higher rates of adverse events during hepatitis C virus therapy in HIV infection: a meta-analysis. J Acquir Immune Defic Syndr. 2010 Oct;55(2):170-5. doi: 10.1097/QAI.0b013e3181e36420. PMID 20622678